CLINICAL TRIAL: NCT02682693
Title: Investigating Denosumab as an add-on Neoadjuvant Treatment for RANK-positive or RANK-negative Primary Breast Cancer and Two Different Nab-Paclitaxel Schedules ; 2x2 Factorial Design (GeparX)
Brief Title: Denosumab as an add-on Neoadjuvant Treatment (GeparX)
Acronym: GeparX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Amgen (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GBG 88
Record Dates: First submitted 2016-01-27; First posted 2016-02-15 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer Female NOS; Tubular Breast Cancer Stage II; Mucinous Breast Cancer Stage II; Invasive Ductal Breast Cancer; HER2 Positive Breast Cancer; Inflammatory Breast Cancer; Tubular Breast Cancer Stage III
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Inflammatory Breast Neoplasms | interventions — Denosumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Epirubicin; Cyclophosphamide; Carboplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Denosumab (Experimental): Denosumab every 4 weeks for 6 cycles.
  Interventions: Drug: Denosumab
- nab-Paclitaxel weekly (Experimental): nab-Paclitaxel weekly for 12 weeks. Patients with HER2-positive tumors receive Trastuzumab and Pertuzumab. Patients with triple-negative tumors receive Carboplatin in parallel to nab-paclitaxel.
  Interventions: Drug: nab-Paclitaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- nab-paclitaxel 2 of 3 weeks (Experimental): nab-Paclitaxel day 1,8 q22 for 12 weeks. Patients with HER2-positive tumors receive Trastuzumab and Pertuzumab. Patients with triple-negative tumors receive Carboplatin weekly in parallel to nab-paclitaxel.
  Interventions: Drug: nab-Paclitaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- EC every two weeks or every three weeks (Experimental): Epirubicin and Cyclophosphamide 600mg/m² for 4 times. Patients with HER2-positive tumors receive Trastuzumab and Pertuzumab.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Denosumab — Denosumab 120 mg every 4 weeks for 6 cycles
  Other Names: Human monoclonal IgG2 antibody
  Arms: Denosumab
Drug: nab-Paclitaxel — nab-paclitaxel 125 mg/m² weekly for 12 weeks or at day 1,8 q22 for 4 cycles (12 weeks)
  Other Names: Abraxane
  Arms: nab-Paclitaxel weekly; nab-paclitaxel 2 of 3 weeks
Drug: Epirubicin — Epirubicin 90 mg/m² every 2 or 3 weeks for 4 times
  Other Names: Farmorubicin
  Arms: EC every two weeks or every three weeks
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m² every 2 or 3 weeks for 4 times
  Other Names: Endoxan
  Arms: EC every two weeks or every three weeks
Drug: Carboplatin — Carboplatin AUC 2 weekly in parallel to nab-Paclitaxel
  Other Names: Diamminplatin(II)-cyclobutan-1,1-dicarboxylat
  Arms: nab-Paclitaxel weekly; nab-paclitaxel 2 of 3 weeks
Drug: Trastuzumab — Trastuzumab 6 (8) mg/kg every 3 weeks simultaneously to all chemotherapy cycles
  Other Names: Herceptin
  Arms: EC every two weeks or every three weeks; nab-Paclitaxel weekly; nab-paclitaxel 2 of 3 weeks
Drug: Pertuzumab — Pertuzumab 420 (840) mg every 3 weeks simultaneously to all chemotherapy cycles
  Other Names: Perjeta
  Arms: EC every two weeks or every three weeks; nab-Paclitaxel weekly; nab-paclitaxel 2 of 3 weeks

SUMMARY:
Pharmacologic inhibition of RANKL attenuates the development of mammary carcinoma and inhibits metastatic progression in multiple mouse models.

In a retrospective analysis it could be demonstrated that elevated expression of RANK was found in 14.5% of patients overall, with a significant predominance in patients with hormone-receptor-negative disease. Expression of RANK was associated with a higher pathological complete response rate but with a shorter disease-free and overall survival. The ABCSG-18 study showed that adjuvant denosumab reduces clinical fractures, improves bone health, and can be administered without added toxicity.

It appears therefore reasonable to test denosumab, a clinically available antibody against RANKL in patients with hormone-receptor-negative primary breast cancer as an adjunct to neoadjuvant chemotherapy for its ability to increase pCR rate and improve outcome in relation to the expression of RANK.

DETAILED DESCRIPTION:
RANK ligand (RANKL), a key factor for bone remodeling and metastasis, is crucial for the development of mouse mammary glands during pregnancy. RANKL functions as a major paracrine effector of the mitogenic action of progesterone in mouse and human mammary epithelium via its receptor RANK and has a role in ovarian hormone-dependent expansion and regenerative potential of mammary stem cells. Pharmacologic inhibition of RANKL attenuates the development of mammary carcinoma and inhibits metastatic progression in multiple mouse models.

In a retrospective analysis of 601 patients treated in the GeparTrio study with chemotherapy (TAC) it could be demonstrated that elevated expression of RANK (immunohistochemical score > 8.5 using the N-1H8 antibody by Amgen) was found in 14.5% of patients overall, with a significant predominance in patients with hormone-receptor-negative disease (33.7% vs 6.4% tumors positive for RANK). Expression of RANK was associated with a higher pathological complete response rate (pCR) (23.0% vs 12.6%) but with a shorter disease-free and overall survival. The ABCSG-18 study showed that adjuvant denosumab reduces clinical fractures, improves bone health, and can be administered without added toxicity. Moreover denosumab improves disease-free survival in postmenopausal woman with hormone receptor positive breast cancer.

It appears therefore reasonable to test denosumab, a clinically available antibody against RANKL in patients with hormone-receptor-negative primary breast cancer as an adjunct to neoadjuvant chemotherapy for its ability to increase pCR rate and improve outcome in relation to the expression of RANK.

ELIGIBILITY:
Inclusion criteria:

* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration from the breast lesion alone is not sufficient. Incisional biopsy or axillary clearance is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Tumor lesion in the breast with a palpable size of 2 cm or a sonographical size of 1 cm in maximum diameter. The lesion has to be measurable in two dimensions, preferably by sonography. In case tumor isn't measurable by sonography, then MRI or mammography is sufficient. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
* Patients must have stage cT1c - cT4a-d disease.
* In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.
* Centrally confirmed ER-negative and PR-negative status. Central pathology includes also assessment of HER2, Ki-67, TIL and RANK status on core biopsy. ER/PR negative is defined as ≤1% stained cells and HER2-positive is defined as IHC 3+ or in-situ hybridization (ISH) and according to ASCO-CAP guidelines as of 2013. LPBC (lymphocyte predominant breast cancer) is defined as more than 50% stromal tumour infiltrating lymphocytes. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy has therefore to be sent to the GBG central pathology laboratory prior to randomization.

Exclusion criteria:

* Patients with stages cT1a, cT1b, or any M1.
* Prior chemotherapy for any malignancy.
* Prior radiation therapy for breast cancer.
* History of disease with influence on bone metabolism, such as osteoporosis, Paget's disease of bone, primary hyperparathyroidism requiring treatment at the time of randomization or considered likely to become necessary within the subsequent six months.
* Use of bisphosphonates or denosumab within the past 1 year.
* Significant dental/oral disease, including prior history or current evidence of osteonecrosis/ osteomyelitis of the jaw, active dental or jaw condition which requires oral surgery, non-healed dental/oral surgery, planned invasive dental procedure for the course of the study.
* Previous malignant disease being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
* Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP >140 / 90 mm Hg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* Currently active infection.
* Incomplete wound healing.
* Definite contraindications for the use of corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
pcR rates of neoadjuvant treatment with or without denosumab in addition to nab-paclitaxel and EC. | 24 weeks
pcR (ypT0 ypN0) rates of nab-Paclitaxel weekly for 12 weeks or 2 of 3 weeks for 12 weeks | 12 weeks

SECONDARY OUTCOMES:
To test for interaction of denosumab treatment with RANK expression. | 24 weeks
To assess the pCR rates per arm for both randomizations separately for TNBC and HR-/HER2+ tumors. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Uwe Blohmer, MD, Principal Investigator — Charite Campus Mitte
Locations (1):
- Charité Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Blohmer JU, Link T, Reinisch M, Just M, Untch M, Stotzer O, Fasching PA, Schneeweiss A, Wimberger P, Seiler S, Huober J, Thill M, Jackisch C, Rhiem K, Solbach C, Hanusch C, Seither F, Denkert C, Engels K, Nekljudova V, Loibl S; GBG and AGO-B. Effect of Denosumab Added to 2 Different nab-Paclitaxel Regimens as Neoadjuvant Therapy in Patients With Primary Breast Cancer: The GeparX 2 x 2 Randomized Clinical Trial. JAMA Oncol. 2022 Jul 1;8(7):1010-1018. doi: 10.1001/jamaoncol.2022.1059. PMID 35588050
- [Derived] Denkert C, Seither F, Schneeweiss A, Link T, Blohmer JU, Just M, Wimberger P, Forberger A, Tesch H, Jackisch C, Schmatloch S, Reinisch M, Solomayer EF, Schmitt WD, Hanusch C, Fasching PA, Lubbe K, Solbach C, Huober J, Rhiem K, Marme F, Reimer T, Schmidt M, Sinn BV, Janni W, Stickeler E, Michel L, Stotzer O, Hahnen E, Furlanetto J, Seiler S, Nekljudova V, Untch M, Loibl S. Clinical and molecular characteristics of HER2-low-positive breast cancer: pooled analysis of individual patient data from four prospective, neoadjuvant clinical trials. Lancet Oncol. 2021 Aug;22(8):1151-1161. doi: 10.1016/S1470-2045(21)00301-6. Epub 2021 Jul 9. PMID 34252375